CLINICAL TRIAL: NCT03476265
Title: Evaluation of Gastroesophageal Reflux Disease - Health Related Quality of Life After Lower Esophageal Sphincter (LES) Stimulation in Patients With Ineffective Esophageal Motilitygus (IEM)
Brief Title: Lower Esophageal Sphincter (LES) Stimulation in Patients With Ineffective Esophageal Motility
Acronym: DYSMOSTIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Austrian Society Of Surgical Oncology (Other)
Responsible Party: Principal Investigator, Matthias Paireder, Consultant at the Division of Surgery at the Medical University of Vienna, Austrian Society Of Surgical Oncology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AUT-DYSMOSTIM-01
Record Dates: First submitted 2018-03-13; First posted 2018-03-26 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Quality of Life; Dysphagia; Electrical Stimulation of the Lower Esophageal Sphincter; Gastro Esophageal Reflux
MeSH Terms: conditions — Deglutition Disorders; Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ineffective Esophageal Motility and GERD (Experimental): Patients with gastroesophageal reflux disease (GERD) refractory to proton pump inhibitors (PPI) and ineffective esophageal motility (IEM) according to the Chicago classification v3.0.
  Interventions: Device: Electrical Stimulation of the Lower Esophageal Sphincter

INTERVENTIONS:
Device: Electrical Stimulation of the Lower Esophageal Sphincter — Laparoscopic implantation of an electrical stimulation device to perform an electrical sphincter augmentation for the treatment of GERD.

SUMMARY:
The aim of this study is to evaluate gastroesophageal reflux disease - health related quality of life (GERD-HRQL) after electrical stimulation of the lower esophageal sphincter (LES) in patients with gastroesophageal reflux disease (GERD) and esophageal dysmotility.

DETAILED DESCRIPTION:
Background The growing burden of gastroesophageal reflux disease (GERD) still impacts healthcare costs intensively. Although the treatment with proton pump inhibitor (PPI) is effective in many cases, surgical treatment remains relevant due to a large amount of PPI refractory GERD. Laparoscopic fundoplication (LF) is considered as standard procedure, but this type of surgery is linked to side effects as dysphagia, gas bloating and inability to belch. Especially patients with ineffective esophageal motility (IEM) are prone to postoperative dysphagia after LF. Lower esophageal sphincter electrical stimulation (LES-EST) was introduced as an alternative technique to avoid side effects of LF. Rodriquez et al. have bee demonstrated that LES-EST significantly raises the LES pressure and improved GERD symptoms such as heartburn and regurgitation. The advantage of this procedure is that the anatomy of the esophageal-gastric junction is not altered dramatically. Notably, patients with severely disordered esophageal peristalsis will benefit from this low-risk profile.

After successful implementation of this technique at the Medical University of Vienna (EK 1149/2014), a prospective evaluation of data with the well established gastroesophageal reflux disease - health-related quality of life is next. Patients with esophageal motility disorder, who undergo LES-EST, will be investigated towards side effects such as gas-bloating, inability to belch, flatulence and dysphagia.

ELIGIBILITY:
Inclusion Criteria:

* Subject is indicated for LES Stimulation and plans to undergo antireflux surgery.
* Subject is meeting the criteria of IEM (Chicago classification v3.0)
* Subject provides signed informed consent

Exclusion Criteria:

* Subject is within a vulnerable population or is unable to understand the informed consent.
* Subject is unwilling to attend follow-up visits.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-01-15 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
Change in patient's GERD-HRQL from baseline to 6 months. | 6 months
  GERD related quality of life (QoL) is assessed with the "gastroesophageal reflux disease - health related quality of life" (GERD-HRQL) questionnaire. QoL is measured at baseline and at six months afters surgery. At unscheduled follow up visits QoL assessment is non-compulsory. The GERD-HRQL score consists of ten questions regarding GERD-related symptoms and their influence on QoL. Total scores range from 0 to 75. Testing will be split to a questionnaire for heartburn (0-30) and a questionnaire for regurgitation (0-30), the two cardinal symptoms of GERD. Lower scores indicate better QoL. This questionnaire was designed to objectively quantify symptom severity and was described validated by Velanovich et al and since then is the most frequently used GERD specific questionnaire.

SECONDARY OUTCOMES:
Change of pH-metry from baseline to 6 months follow up | 6 months
  Total % of time of pH < 4 in 24 hours impedance/pH reflux monitoring (ZepHr®, Sandhill Scientific Inc., USA).
Change of number of reflux events >1minute and >5 minute duration from baseline to 6 months follow up | 6 months
  24 hours impedance/pH reflux monitoring (ZepHr®, Sandhill Scientific Inc., USA).
Distal Contractile Integral | 6 months
  High-resolution impedance manometry (InSIGHT Ultima®, Sandhill Scientific Inc., USA)

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian F Schoppmann, MD, Study Director — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Peery AF, Crockett SD, Barritt AS, Dellon ES, Eluri S, Gangarosa LM, Jensen ET, Lund JL, Pasricha S, Runge T, Schmidt M, Shaheen NJ, Sandler RS. Burden of Gastrointestinal, Liver, and Pancreatic Diseases in the United States. Gastroenterology. 2015 Dec;149(7):1731-1741.e3. doi: 10.1053/j.gastro.2015.08.045. Epub 2015 Aug 29. PMID 26327134
- [Background] Subramanian CR, Triadafilopoulos G. Refractory gastroesophageal reflux disease. Gastroenterol Rep (Oxf). 2015 Feb;3(1):41-53. doi: 10.1093/gastro/gou061. Epub 2014 Sep 30. PMID 25274499
- [Background] Richter JE. Gastroesophageal reflux disease treatment: side effects and complications of fundoplication. Clin Gastroenterol Hepatol. 2013 May;11(5):465-71; quiz e39. doi: 10.1016/j.cgh.2012.12.006. Epub 2012 Dec 23. PMID 23267868
- [Background] Novitsky YW, Wong J, Kercher KW, Litwin DE, Swanstrom LL, Heniford BT. Severely disordered esophageal peristalsis is not a contraindication to laparoscopic Nissen fundoplication. Surg Endosc. 2007 Jun;21(6):950-4. doi: 10.1007/s00464-006-9126-3. Epub 2006 Dec 20. PMID 17177077
- [Background] Rodriguez L, Rodriguez P, Neto MG, Ayala JC, Saba J, Berel D, Conklin J, Soffer E. Short-term electrical stimulation of the lower esophageal sphincter increases sphincter pressure in patients with gastroesophageal reflux disease. Neurogastroenterol Motil. 2012 May;24(5):446-50, e213. doi: 10.1111/j.1365-2982.2012.01878.x. Epub 2012 Jan 31. PMID 22292889
- [Background] Rodriguez L, Rodriguez PA, Gomez B, Netto MG, Crowell MD, Soffer E. Electrical stimulation therapy of the lower esophageal sphincter is successful in treating GERD: long-term 3-year results. Surg Endosc. 2016 Jul;30(7):2666-72. doi: 10.1007/s00464-015-4539-5. Epub 2015 Oct 20. PMID 26487200
- [Background] Velanovich V. The development of the GERD-HRQL symptom severity instrument. Dis Esophagus. 2007;20(2):130-4. doi: 10.1111/j.1442-2050.2007.00658.x. PMID 17439596
- [Background] Velanovich V. Comparison of generic (SF-36) vs. disease-specific (GERD-HRQL) quality-of-life scales for gastroesophageal reflux disease. J Gastrointest Surg. 1998 Mar-Apr;2(2):141-5. doi: 10.1016/s1091-255x(98)80004-8. PMID 9834409
- [Derived] Paireder M, Kristo I, Asari R, Jomrich G, Steindl J, Rieder E, Schoppmann SF. Effect of electrical stimulation therapy of the lower esophageal sphincter in GERD patients with ineffective esophageal motility. Surg Endosc. 2021 Nov;35(11):6101-6107. doi: 10.1007/s00464-020-08104-3. Epub 2020 Oct 30. PMID 33128080